CLINICAL TRIAL: NCT02152202
Title: Does a Semi-upright Position During Sleep Prevent Worsening of Severity of Obstructive Sleep Apnea (OSA) on the Second Postoperative Night in Patients Following Elective Inpatient Surgery? A Two Arm, Parallel, Randomized, Controlled, First Stage Proof of Concept Trial
Brief Title: Semi-up Right Position Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Staff Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol version july 17, 2011
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Supine Position; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semi-upright position (Experimental): Semi-upright position defined as 45 degrees incline from horizontal of the patients bed during nocturnal sleep, for two postoperative nights. Daytime naps will be excluded. A regular pillow may be used by the patients based upon the level of comfort and also to support the head in a neutral position.
  Interventions: Other: Semi-upright position
- Control group (Supine position) (Other): In this group patients' bed will be set into Supine/0 degree angle during sleep in the night time. Patient will be managed according to routine care
  Interventions: Other: Supine position

INTERVENTIONS:
Other: Semi-upright position — In this group patients' bed will be set into 45 degree angle during sleep in the night time.
  Other Names: Semi-upright position (45 degree bed angle)
  Arms: Semi-upright position
Other: Supine position — Control: Supine position during nocturnal sleep for at least two postoperative nights.
  Other Names: Control group
  Arms: Control group (Supine position)

SUMMARY:
Our main objective is to perform an explanatory, first stage proof of concept, randomized controlled trial to determine whether a semi-upright patient position versus a supine position while asleep in the postoperative period helps decrease the worsening of AHI in patients diagnosed with OSA and compare this to usual care (i.e. supine patient positioning while asleep).

The investigators will evaluate whether a semi-upright position reduces: worsening of AHI (as measured with a portable PSG) on the second postoperative night (POD2); oxygen desaturation index (using a portable oxygen saturation monitor, oxygen desaturation defined as >4% change below baseline lasting for 10 seconds); REM sleep related change in AHI at baseline and POD2.; major and minor perioperative complications on postoperative day POD1, POD2, at discharge and POD 30.; length of hospital stay and readmission within 30 days; and patient satisfaction score on POD30

DETAILED DESCRIPTION:
The proposed study is to determine whether patient positioning in supine or semi-sitting position can effectively control the worsening of OSA see in the postoperative period.

The study patient will be randomized to semi-sitting position (45 degrees incline) group or supine (0 degrees incline) group. Patients will undergo a portable sleep study on the first or second postoperative night. They will also be monitored with wristwatch oximeter pre and postoperatively according to the study protocol. Patients will be managed according to the routine care determined by the health care team. There will be no change in the clinical management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and above),
* ASA physical status I to IV,
* Undergoing elective inpatient surgery with obstructive sleep apnea (as determined by initial screening using STOP-Bang questionnaire and if at high risk (>3 points),
* Confirmed by an Apnea-hypopnea index (AHI) >5 using a diagnostic home portable polysomnography)

Exclusion Criteria:

* Patients previously diagnosed as OSA and on continuous positive airway pressure (CPAP) device;
* Known cervical, shoulder, spine abnormalities, and/or chronic pain predisposing to difficulty in maintaining a sitting position; or
* Previous intervention for OSA (e.g., uvulopalatopharyngoplasty, bariatric surgery); where sitting position is contraindicated postoperatively such as hip or spine surgery, hemodynamic instability; ambulatory surgery i.e. planned discharge on the same day of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Comparison of worsening of severity of OSA using the Apnea-hypopnea index (AHI) as determined by a portable polysomnography study from baseline (preoperatively) to the second postoperative night. | 3days
  The AHI is used as a surrogate outcome to establish the diagnosis of OSA (AHI>5) and severity of OSA as per the guidelines from American Academy of Sleep Physicians (AASP).5 It is a continuous outcome and is measured by counting the number of apneas (complete cessation of airflow for more than 10 s) and hypopneas (airflow reduction more than 50%) despite continuing breathing efforts and thus differentiating from central events (absence of breathing efforts). The relationship of AHI to clinical outcomes of relevance has been well established in the literature.

SECONDARY OUTCOMES:
Major and minor perioperative complications and length of hospital stay on postoperative day (POD) 1, POD2, at discharge and POD 30 will be recorded based on chart review. | 30 days
  The oxygen desaturation index; REM sleep related change in AHI at baseline and POD2 and time spent in lateral position while asleep will be deciphered from the PSG data.
Hospital stay | 30 days
  Length of hospital stay, readmission within 30 days, and patient satisfaction score will be recorded and telephonic interview with the patient on POD30.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Department of Anesthesia, Toronto, Ontario
  - Toronto Western Hospital, Department of Aneshtesia, Toronto, Ontario
  - University Health Network, Department of Anesthesia, Toronto, Ontario

REFERENCES:
- [Derived] Lukachan GA, Yadollahi A, Auckley D, Gavrilovic B, Matelski J, Chung F, Singh M. The impact of semi-upright position on severity of sleep disordered breathing in patients with obstructive sleep apnea: a two-arm, prospective, randomized controlled trial. BMC Anesthesiol. 2023 Jul 13;23(1):236. doi: 10.1186/s12871-023-02193-y. PMID 37443016